CLINICAL TRIAL: NCT03864718
Title: Efficacy of Photodynamic Therapy and Intra-lesional 5-wing in Complex Perianal Fistula
Brief Title: Photodynamic Therapy in Anal Fistula
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Antonio Arroyo Sebastian, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: TFD-ALA
Record Dates: First submitted 2019-03-03; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Rectal Fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Photochemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- complex anal fistula
  Interventions: Procedure: photodynamic therapy

INTERVENTIONS:
Procedure: photodynamic therapy — Intralesional 5-aminolevulinic acid gel 2% was directly injected into the fistula. The internal and external orifices were closed. After an incubation period of 2 h, the fistula was irradiated using an optical fibre connected to a red laser (MULTIDIODE 630 PDT, INTERmedic, Spain) operating at 1 W/ cm for 3 min (180 Joules).

SUMMARY:
Objective: Validate and analyze the results of intralesional photodynamic therapy in the treatment of complex anal fistula.

Methods: Prospective observational study including patients treated for complex anal fistula who underwent intralesional photodynamic therapy (i-PDT). Patients were included with a minimum follow up of 1-year, in order to evaluate recurrence, continence and postoperative morbidity. Intralesional 5-aminolevulinic acid gel 2% was directly injected into the fistula. The internal and external orifices were closed. After an incubation period of 2 h, the fistula was irradiated using an optical fibre connected to a red laser (MULTIDIODE 630 PDT, INTERmedic, Spain) operating at 1 W/ cm for 3 min (180 Joules).

ELIGIBILITY:
Inclusion Criteria:

* complex anal fistula according to Parks classification

Exclusion Criteria:

* Non cryptoglandular fistulas
* acute sepsis
* inflammatory bowel diseases
* simple fistulas (defined as subcutaneous, intersphincteric and low transsphincteric fistula)
* pregnant patients
* ASA IV
* patients <18
* immunocompromised
* patients who refused consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Healing | 12 months after surgery
  Yes/Not